CLINICAL TRIAL: NCT02828449
Title: Assessment of the Implementation of a Therapeutic Educational Intervention Affecting Adherence to Oral Chemotherapy
Brief Title: Assesment of the Implementation of a Therapeutic Educational Intervention Affecting Adherence to Oral Chemotherapy
Acronym: CHIMIO ORALE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Cancérologie de la Loire (Other)
Collaborators: Hospices Civils de Lyon (Other); Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-12
Record Dates: First submitted 2016-02-25; First posted 2016-07-11 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- therapeutic education program (Experimental): therapeutic education program which aims is to improve the adherence to the treatment and management of adverse effects of this treatment in patients taking an oral chemotherapy for active cancer
  Interventions: Behavioral: therapeutic education program

INTERVENTIONS:
Behavioral: therapeutic education program

SUMMARY:
Therapeutic education is an effective way to support the prescription of oral chemotherapy in oncology. It aims to increase adherence to treatment, to better control the side effects and reduce unplanned readmissions. The three major oncology institutions in the Rhône-Alpes region (Hospices Civils de Lyon, the Centre Léon Bérard Cancer Institute and Lucien Neuwirth) decided to collaborate on a project to implement an adapted Therapeutic Education Program context of each of these institutions.

The objective of this study is to evaluate the implementation of the intervention in the 3 participating centers, over 1 year:

1. Assess the achievement of the target population
2. Evaluate the adaptation of intervention in context
3. Evaluate the effectiveness of the intervention (impact): effectiveness in real life, identification of interactions with the environment linked to the center, identification of unintended effects of the intervention.
4. Assessing the sustainability of the intervention

ELIGIBILITY:
Inclusion Criteria:

* Patient care in medical oncology services of the Cancer Institute of Lucien Neuwirth, the Lyon-Sud hospital and the Centre Léon Bérard:
* Age over 18 years
* Introducing an active cancer (local extension, locoregional or metastatic)
* Oral chemotherapy as monotherapy or in combination with other treatments, initiated or in progress

Exclusion Criteria:

* Refusal to participate, protected adult patient under guardianship.
* Patient disability to understand the course of the study, the Therapeutic education program, or failure to follow the educational sessions.
* Patient with documented history of cognitive or psychiatric disorders.
* Patient on adjuvant therapy or hormone therapy for prostate cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
percentage of affected population | 3 months
Level of acquisition of knowledge | 3 months
  Questionnaire composed of numerous questions dealing with patient's knowledge about his/her disease, treatment and treatment's side effects . Answers are quoted in Yes/No and a global scoring is made with all answers. Final measure is a percentage of good answers.
Anxiety and Depression | 3 months
  measured with the Hospital Anxiety Depression Scale (Zigmond & Snaith, 1983 ), wich gives separated results about the level of anxiety and of depression according to the level of scoring to a set of 14 questions. Questions are rated from 0-3, and the anxiety and depression subscale scores range from 0-21. The cutoff for each subscale is eight.
Quality of Life Questionnaire | 3 months
Morisky Measurement Adherence Scale | 3 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Léon Bérard, Lyon
  - CH Lyon Sud, Pierre-Bénite
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No